CLINICAL TRIAL: NCT04149587
Title: A Canadian Phase IV, Multicenter, Single-Arm Study To Evaluate the Effectiveness of Treatment With Brodalumab (SILIQ) in Psoriasis Patients With Inadequate Response to Their Current Biologic Agent Regimen
Brief Title: A Study of Brodalumab (SILIQ®) in Psoriasis Participants With Inadequate Response to Their Current Biologic Agent Regimen
Status: Completed | Type: Observational
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BHS-CAN-DERM-002
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — brodalumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Brodalumab 210 mg Q2W: Participants will receive brodalumab 210 milligrams (mg) administered as 1 subcutaneous injection at Day 1 and at Weeks 1 and 2 followed by 210 mg every 2 weeks (Q2W) thereafter until Week 26.
  Interventions: Drug: Brodalumab

INTERVENTIONS:
Drug: Brodalumab — Brodalumab will be administered per dose and schedule specified in the arm.
  Other Names: SILIQ®

SUMMARY:
This multicenter, prospective, observational, single-arm, 26-week study will evaluate the effectiveness, safety and tolerability of brodalumab subcutaneous injection in participants with psoriasis with inadequate response to their current biologic agent regimen.

ELIGIBILITY:
Inclusion Criteria:

* Participant has enrolled in the brodalumab patient support program (PSP).
* Participant has provided informed consent, using an Independent Ethics Committee (IEC) or Institutional Review Board (IRB) approved Informed Consent Form (ICF).
* Confirmed diagnosis with moderate to severe plaque psoriasis.
* On stable treatment with a biologic for a minimum of 12 weeks, and not having achieved adequate therapeutic response, as per the investigator's judgment, for example BSA of greater than or equal to (≥) 1% and physicians global assessment (PGA) of ≥3.
* Participant must be able to understand and communicate with the investigator, as well as complete the study questionnaires, in one of the available and validated languages.
* Participants participating in other observational studies or registries are permitted to enroll in this study at the same time.

Exclusion Criteria:

* Receiving or has received any investigational drug (or is currently using an investigational device) within 30 days or 5 drug half-lives (whichever is longer) prior to receiving the first dose of brodalumab (Day 1).
* Participant has a history of any psychiatric disorder or substance abuse that, in the opinion of the investigator, would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion.
* Participant has previous history of suicidal ideation and/or behavior or report suicidal ideation and/or behavior during the study.
* Presence of any other serious and/or uncontrolled medical condition that, in the opinion of the investigator, prohibits the participant from participating in the study.
* Participant has a body mass index (BMI) greater than (>) 40 kilograms/square meter (kg/m^2) during the screening phase or during the study.
* Any contraindication as per the product monograph: Brodalumab injection is contraindicated in participants with clinically significant hypersensitivity to brodalumab or to any of the excipients or component of the container. Brodalumab is contraindicated in participants with Crohn's disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who did not respond adequately to treatment with their current biological regimen as per the investigator clinical judgement
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Psoriasis Area and Severity Score (PASI) 100 Response at Week 26 | Week 26
  PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72(maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4). PASI 100 responders were defined as participants achieving 100% improvement at Week 26.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Static Physicians Global Assessment (sPGA) Score 0/1 | Weeks 1, 2, 4, 16, and 26
  The sPGA scale (0 [clear] to 4 [severe]) will be completed by the investigator or qualified designee and is designed to evaluate the assessor's global assessment of the participant's psoriasis. 0 (clear) = No signs of psoriasis; postinflammatory hyperpigmentation may be present, 1 (almost clear) = No thickening; normal to pink coloration; no to minimal focal scaling, 2 (mild) = Just detectable to mild thickening; pink to light red coloration; predominantly fine scaling, 3 (moderate) = Clearly distinguishable to moderate thickening; dull to bright red, moderate scaling, 4 (severe) = Severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions.
Change From Baseline in Mean sPGA * Body Surface Area (BSA) Score at Weeks 1, 2, 4, 16, and 26 | Baseline, Weeks 1, 2, 4, 16, and 26
  The area of body surface affected by psoriasis will be estimated by the investigator as a percentage of the participant's total BSA wherein the area of the participant's palm will be considered as 1% of total BSA. sPGA of disease severity is measured by the investigator on a 6-point scale wherein 0=Clear, 1=Almost Clear, 2=Mild, 3=Moderate, 4=Severe, 5=Very Severe. The product of these values offers a more specific assessment of the severity of psoriasis. This product can yield a result between 0 (no disease) and 500 (most severe disease).
Percentage of Participants Achieving PASI 75 and PASI 90 | Weeks 1, 2, 4, 16, and 26
  PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72(maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4). PASI 75 responders were defined as participants achieving ≥75% improvement at specified timepoints. PASI 90 responders were defined as participants achieving ≥90% improvement at specified timepoints.
Percentage of Participants Achieving PASI 100 at Weeks 1, 2, 4, and 16 | Weeks 1, 2, 4, and 16
  PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72(maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4). PASI 100 responders were defined as participants achieving 100% improvement at specified timepoints.
Change From Baseline in Psoriasis Symptoms Inventory (PSI) Score at Weeks 1, 2, 4, 16, and 26 | Baseline, Weeks 1, 2, 4, 16, and 26
  The PSI is a psoriasis-specific patient-reported outcome that measures the severity of psoriasis signs and symptoms based on an 8-item scale. The severity of itch, redness, scaling, burning, stinging, cracking, flaking, and pain over the last 24 hours is assessed on a scale of 0 to 4 (not at all, mild, moderate, severe, or very severe) for a total score of 32, with higher scores indicating more severe disease.
Change From Baseline in Dermatology Life Quality Index (DLQI) Score at Weeks 1, 2, 4, 16, and 26 | Baseline, Weeks 1, 2, 4, 16, and 26
  The DLQI is a 10-item general dermatology disability index designed to assess health-related quality of life in adult participants with skin conditions. The measure is self-administered and includes domains of daily activities, leisure, personal relationships, symptoms and feelings, treatment, and work/school. Each item has four response categories, ranging from 0 (not at all or not relevant) to 3 (very much) assessing the impact of the disease over the last week. The DLQI total score is a sum of the 10 questions. Scores range from 0 to 30 and higher scores indicate greater health-related quality-of-life impairment.
Change From Baseline in Hospital Anxiety and Depression Scale (HADS) Score at Weeks 1, 2, 4, 16, and 26 | Baseline, Weeks 1, 2, 4, 16, and 26
  The HADS is a self-reported questionnaire that assesses anxiety and depression. The scale includes two subscales, specifically depression and anxiety. Each subscale has 7 items, for a total of 14 items with a total score ranging from 0 to 21 for each scale. Participants report the relative frequency of symptoms over the past week using a 4-point Likert scale ranging from 0 to 3. Higher scores indicate a greater likelihood of depression or anxiety.
Change From Baseline in EuroQoL-5 Dimensional (EQ-5D) With Psoriasis Bolt-on (EQ-PSO) Score at Weeks 1, 2, 4, 16, and 26 | Baseline, Weeks 1, 2, 4, 16, and 26
  The EQ-PSO is a psoriasis-specific adaptation of the EQ-5D, a standardized measure of health status that can be used to provide a simple, generic measure of health outcome. The EQ-5D comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each of which is assessed by the respondent according to 5 levels (no problems, slight problems, moderate problems, severe problems, and extreme problems.). The EQ-PSO includes two additional, psoriasis-specific dimensions: skin irritation and self-confidence.
Number of Participants With Adverse Events (AEs) | Baseline (Week 0) up to end of treatment (Week 26)
Time to Onset of Action | Baseline up to Week 26
Number of Participants Adhering to the Treatment | Baseline up to Week 26
Percentage of Participants Achieving PASI 75, PASI 90, and PASI 100 at Week 16 and 26 According to the Last Biologic Agent That the Participant was Receiving Before Initiating Treatment With Brodalumab | Week 16 and 26
  PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72(maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4). PASI 75 responders were defined as participants achieving ≥75% improvement at specified timepoints. PASI 90 responders were defined as participants achieving ≥90% improvement at specified timepoints. PASI 100 responders were defined as participants achieving 100% improvement at specified timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Anya Loncaric, Study Director — Bausch Health Americas, Inc.
Locations (11):
- Canada (11):
  - Bausch Site 009, Nanaimo, British Columbia
  - Bausch Site 002, Montréal, Manitoba
  - Bausch Site 001, Winnipeg, Manitoba
  - Bausch Site 007, Markham, Ontario
  - Bausch Site 008, Mississauga, Ontario
  - Bausch Site 014, North Bay, Ontario
  - Bausch Site 005, Ottawa, Ontario
  - Bausch Site 012, Toronto, Ontario
  - Bausch Site 010, Waterloo, Ontario
  - Bausch Site 011, Drummondville, Quebec
  - Bausch Site 003, Surrey, Quebec